CLINICAL TRIAL: NCT04090359
Title: Dual Mobility Acetabular Cups in Revision TJA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Rothman Institute Orthopaedics (Other); Keck School of Medicine of USC (Other); NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17022801
Record Dates: First submitted 2019-09-11; First posted 2019-09-16 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Dislocation, Hip
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two groups: revision THA with dual mobility components vs revision THA with large head, single bearing designs (36mm and 40mm).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Dual Mobility (Experimental): If patients are randomized to the dual mobility cohort, they will receive a dual mobility prosthesis at the surgeon's discretion. All surgeries will be performed via the posterior approach, per the participating surgeon's usual standard. Patients will be on postoperative hip precautions for 6 weeks, per departmental protocol. No braces will be utilized.
  Interventions: Device: Dual Mobility Implant
- Conventional, Single-bearing hip implant (Active Comparator): If patients are randomized to the conventional, single bearing cohort, surgeons will use their preferred implant design at their discretion using a 36 or 40mm head, depending on the diameter of the cup and manufacturer specifications. All surgeries will be performed via the posterior approach, per the participating surgeon's usual standard. Patients will be on postoperative hip precautions for 6 weeks, per departmental protocol. No braces will be utilized.
  Interventions: Device: Conventional, single-bearing implant

INTERVENTIONS:
Device: Dual Mobility Implant — Patients in this intervention will receive a dual mobility implant
  Arms: Dual Mobility
Device: Conventional, single-bearing implant — Patients in this intervention will receive a conventional, single-bearing implant
  Arms: Conventional, Single-bearing hip implant

SUMMARY:
The aim of this study is to the compare clinical outcomes of patients undergoing a revision total hip arthroplasty (THA) with the use of a dual mobility bearing versus a single bearing design with the use of a large femoral head (36mm or 40mm). We hypothesize the use of dual-mobility components in revision THA will be associated with a lower dislocation rate in the first year following surgery.

DETAILED DESCRIPTION:
The aim of this study is to the compare clinical outcomes of patients undergoing a revision total hip arthroplasty (THA) with the use of a dual mobility bearing versus a single bearing design with the use of a large femoral head (36mm or 40mm). We hypothesize the use of dual-mobility components in revision THA will be associated with a lower dislocation rate in the first year following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Any patient older than 18 years of age scheduled for a revision THA, including revision of both components, conversion of a hip resurfacing to THA, conversion of a hemiarthroplasty to THA, and revision of single components which allow implantation of dual-mobility bearings. In addition, patients undergoing reimplantation of a total hip arthroplasty following a two-stage revision for periprosthetic infection will also be included. Only patients with an acetabular shell diameter capable of accommodating at least a 36mm femoral head will be included.

Exclusion Criteria:

* Less than 18 years of age, primary THA,
* conversion of non-arthroplasty femoral neck fracture fixation to THA,
* patients unwilling to participate.
* patients where the surgeon makes the intraoperative decision to use a constrained liner will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2036-12-01 (Estimated)

PRIMARY OUTCOMES:
Prosthetic Dislocation | 6 weeks
  The rate of prosthetic dislocation between the two cohorts will be measured at standard postoperative clinic visits
Prosthetic Dislocation | 3 months
  The rate of prosthetic dislocation between the two cohorts will be measured at standard postoperative clinic visits
Prosthetic Dislocation | 2 years
  The rate of prosthetic dislocation between the two cohorts will be measured at standard postoperative clinic visits
Prosthetic Dislocation | 5 years
  The rate of prosthetic dislocation between the two cohorts will be measured at standard postoperative clinic visits
Prosthetic Dislocation | 10 years
  The rate of prosthetic dislocation between the two cohorts will be measured at standard postoperative clinic visits
Prosthetic Dislocation | 15 years
  The rate of prosthetic dislocation between the two cohorts will be measured at standard postoperative clinic visits
Prosthetic Dislocation | 20 years
  The rate of prosthetic dislocation between the two cohorts will be measured at standard postoperative clinic visits

SECONDARY OUTCOMES:
Complications | up to 20 years after the patient is discharged from the hospital
  Any peri- or postoperative complications will be recorded, including component loosening, occurrence of intraprosthetic dislocation, infection, periprosthetic fractures, revision rates
Routine radiographs assess for loosening and proper component placement | 6 weeks
  Routine radiographs (AP Pelvis, frogleg lateral, and cross-table lateral radiographs) will be obtained at follow-up visits and assessed for cup placement, anteversion, radiographic signs of loosening, and component migration. Radiographics will be assessed for loosening in a yes/no way.
Routine radiographs assess for loosening and proper component placement | 3 months
  Routine radiographs (AP Pelvis, frogleg lateral, and cross-table lateral radiographs) will be obtained at follow-up visits and assessed for cup placement, anteversion, radiographic signs of loosening, and component migration. Radiographics will be assessed for loosening in a yes/no way.
Routine radiographs assess for loosening and proper component placement | 2 years
  Routine radiographs (AP Pelvis, frogleg lateral, and cross-table lateral radiographs) will be obtained at follow-up visits and assessed for cup placement, anteversion, radiographic signs of loosening, and component migration. Radiographics will be assessed for loosening in a yes/no way.
Routine radiographs assess for loosening and proper component placement | 5 years
  Routine radiographs (AP Pelvis, frogleg lateral, and cross-table lateral radiographs) will be obtained at follow-up visits and assessed for cup placement, anteversion, radiographic signs of loosening, and component migration. Radiographics will be assessed for loosening in a yes/no way.
Routine radiographs assess for loosening and proper component placement | 10 years
  Routine radiographs (AP Pelvis, frogleg lateral, and cross-table lateral radiographs) will be obtained at follow-up visits and assessed for cup placement, anteversion, radiographic signs of loosening, and component migration. Radiographics will be assessed for loosening in a yes/no way.
Routine radiographs assess for loosening and proper component placement | 15 years
  Routine radiographs (AP Pelvis, frogleg lateral, and cross-table lateral radiographs) will be obtained at follow-up visits and assessed for cup placement, anteversion, radiographic signs of loosening, and component migration. Radiographics will be assessed for loosening in a yes/no way.
Routine radiographs assess for loosening and proper component placement | 20 years.
  Routine radiographs (AP Pelvis, frogleg lateral, and cross-table lateral radiographs) will be obtained at follow-up visits and assessed for cup placement, anteversion, radiographic signs of loosening, and component migration. Radiographics will be assessed for loosening in a yes/no way.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - New York University Medical Center, New York, New York
  - Rothman Institute, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weintraub MT, DeBenedetti A, Nam D, Darrith B, Baker CM, Waren D, Schwarzkopf R, Courtney PM, Della Valle CJ. Dual-Mobility versus Large Femoral Heads in Revision Total Hip Arthroplasty: Interim Analysis of a Randomized Controlled Trial. J Arthroplasty. 2023 Jul;38(7S):S206-S210. doi: 10.1016/j.arth.2023.03.089. Epub 2023 Apr 3. PMID 37019309